CLINICAL TRIAL: NCT00283829
Title: Immunotherapy With Low Dose Interleukin-2 After Cytoreductive Chemotherapy for Patients With Hormone Refractory Metastatic Prostate Cancer: A Phase I/II Study
Brief Title: Immunotherapy After Chemotherapy for Patients With Hormone Refractory Metastatic Prostate Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Celestia Higano, MD, University of Washington
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 02-3017-A-04; IIT-16117; USI-IL2-01-012
Record Dates: First submitted 2006-01-26; First posted 2006-01-30 (Estimated); Last update posted 2007-11-29 (Estimated); Status verified 2007-11

CONDITIONS: Prostate Cancer
Keywords: Immunotherapy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Docetaxel; Interleukin-2; Interleukins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- I (Other): Docetaxel followed by IL-2
  Interventions: Drug: docetaxel; Drug: IL2

INTERVENTIONS:
Drug: docetaxel — chemotherapy
  Other Names: taxotere
Drug: IL2 — immunotherapy
  Other Names: Interleukin

SUMMARY:
The purpose of this study is to test if interleukin-2, a drug that stimulates the immune system, can be used after chemotherapy to slow the progression of your disease. We also want to test what the best dose of interleukin-2 is that can be used safely at home.

Interleukin-2, abbreviated as IL2, is a naturally produced growth hormone for the immune cells in our body. It stimulates the growth of the immune cells and enhances their ability to fight infections and cancers. In people with cancer, the immune cells are typically suppressed and became even more so after irradiation and chemotherapy treatment. By giving you more IL2 we hope to enhance the immune system so that it can fight the cancer better, control cancer growth and shrink the cancer.

DETAILED DESCRIPTION:
There are two treatment phases in this study. But before you begin in the study, we will need to find out whether you are eligible for the study. You will undergo the following procedures.

* Medical history review and physical exam
* Blood tests for hematology, chemistries, PSA, and immune assays (approximately 4 tablespoons of blood)
* EKG
* CT scan of the abdomen and pelvis and a bone scan
* Complete a pain questionnaire, quality of life questionnaire, pain medication diary, and symptom diary

The initial treatment phase of this study consists of chemotherapy drug given weekly. You will receive 3 weekly chemotherapy treatments followed by 1 week with no treatment. Three weeks of treatment followed by one week of no treatment is considered 1 cycle, and you will receive a total of 4 cycles of chemotherapy over a 16-week period. Taxotere is given intravenously in the clinic on the 1st day of each weekly treatment.

Treatment with taxotere is a currently accepted treatment for this stage prostate cancer. Your doctor may recommend you receive taxotere even if you do not participate in this study. During this phase of treatment, you will have blood draws on treatment weeks prior to having the chemotherapy. You will have a PSA drawn every month (weeks 5, 9, and 13). We will ask you to complete a pain questionnaire, quality of life questionnaire, pain medication diary, and symptom diary at weeks 5, 9, and 13. Some of the questions may be personal, such as "I am satisfied with my sex life" and "I worry about dying". You do not have to answer these questions if you do not want to. You will also have a physical exam at the beginning of your 3rd cycle of treatment (week 9).

The second phase of the treatment program is the experimental part: immunotherapy with IL2. You will be assigned to receive one of 4 doses of IL2. This is because we are testing what is the highest dose of IL2 that a subject can receive without having unacceptable side affects from the IL2. You will give yourself shots of IL2 under the skin twice a day for 5 days per week for 3 weeks. During the 3rd week of treatment there are 2 days when you have to give a higher dose of IL2 for boosting the immune cells (see below diagram). The 4th week will be a rest week where you do not receive treatment. One 4-week period of IL2 treatment is called a cycle. You will continue to receive cycles of IL2 treatment as long as your cancer shows no further growth. We will teach you how to administer the IL2 at home.

ELIGIBILITY:
Inclusion Criteria:

* Patients are age >18 years with histological diagnosis of prostate cancer
* Hormone refractory disease with at least 2 serial rises in PSA with a castrate level of testosterone (< 50ng/dL). Primary hormonal therapy will be continued.
* Patients must have metastatic disease as evidenced by soft tissue or bony metastasis
* Patients have an ECOG performance status of 0, 1, 2
* Patients must have preserved organ function
* Bilirubin < ULN and serum creatinine 1.5 x ULN, transaminases (SGOT and/or SGPT) may be up to 2.5 x institutional upper limit of normal (ULN) if alkaline phosphatase is ULN, or alkaline phosphatase may be up to 4 x ULN if transaminases are ULN.
* Patients must be off chronic steroid treatment for at least 2 weeks, and pre-/post-chemotherapy steroid medication for at least 1 week
* Patients may not receive Taxanes previously.
* Patients must be able to complete pain and quality of life scales.
* Ancillary treatments, such as bisphosphonate, pain medication is allowed, but natural herbal, homeopathic supplements such as MGN-3 is not allowed.
* Absolute neutrophil count > 1,500/mm3, hemoglobin > 8.0 g/dl, platelet count > 100,000/mm3.
* Men of childbearing potential must be willing to consent to using effective contraception while on treatment and for a 12 month period thereafter.

Exclusion Criteria:

* Patients on chronic steroid medication
* Spine radiation therapy for cord compression within 2 weeks of study entry
* Concurrent use of other investigational therapy
* Prior immunotherapy with IL2 or alpha-interferon within 30 days
* Peripheral neuropathy > Grade 1
* Other active malignancy, except non-melanotic skin cancer
* Significant active medical illness or psychosocial condition that in the opinion of the investigator would preclude protocol treatment.
* Hypersensitivity to drugs formulated with polysorbate-80
* Patients with contraindications to Coumadin or aspirin.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2002-09; Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
To determine the feasibility of sequencing low dose SQ IL-2 with chemotherapy in patients with hormone refractory prostate cancer (HRPC) in an outpatient setting. | 2 years

SECONDARY OUTCOMES:
To determine the impact of docetaxel on the natural immune defense system in patients before IL-2 administration. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Celestia Higano, MD, Principal Investigator — University of Washington
Locations (1):
- Seattle Cancer Care Alliance, Seattle, Washington, United States